CLINICAL TRIAL: NCT05068817
Title: Pilates Mat Versus Cervical Stabilization Exercises on Craniovertebral Angle, Pain, Function of Daily Life, Cervical Range of Motion, Dynamic Balance in Young Adults With Forward Head Posture: Randomized Controlled Trial
Brief Title: Pilates Mat Versus Cervical Stabilization Exercises on Balance in Young Adults With Forward Head Posture
Acronym: FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, Doctor of physical therapy, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/003348
Record Dates: First submitted 2021-09-16; First posted 2021-10-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Musculoskeletal Diseases
Keywords: Balance; Craniovertebral angle
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates mat exercises (Experimental): one hour Pilates exercises with 10 min warm up and 5-10 min cooling down
  Interventions: Other: Pilates mat exercises; Other: conventional physiotherapy
- cervical stabilization exercises (Experimental): training of deep cervical flexor muscles with pressure biofeedback unit
  Interventions: Other: cervical stabilization exercises; Other: conventional physiotherapy
- conventional physiotherapy (Active Comparator): 10 min hot pack on cervical area range of motion exercises and isometric neck exercises as a home program
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Pilates mat exercises — Pilates mat exercises: Each Pilates session will last for one hour and commence with a 10 minute warm up and finish with a 10 min cool down. The subjects will be taught the 5 key elements of Pilates (lateral costal breathing, centring which is a neutral position of the lumbar spine with activation of the core muscles, ribcage placement, shoulder blade placement and neutral position of the cervical spine with slight upper cervical flexion at the cranio-cervical junction).
  Pilates exercise program will consist of warm up exercises, main treatment program (10 level) and cooling down exercises.
  Arms: Pilates mat exercises
Other: cervical stabilization exercises — training of deep cervical flexor muscles with pressure biofeedback unit, 20 min/day, 3 days/week for 12 weeks.
  Arms: cervical stabilization exercises
Other: conventional physiotherapy — 10 min hot pack on cervical area range of motion exercises and isometric neck exercises as a home program 3 days/week for 12 weeks

SUMMARY:
see if there will be no statistical significant difference between the effects of Pilates mat versus cervical stabilization exercises on dynamic balance in young adults with forward head posture.

DETAILED DESCRIPTION:
In modernized time, extended use of mobile phone and computers has increased anterior weight bearing of cervical spine leading to a variety of musculoskeletal disorders related to the neck by changing the biomechanical stress of cervical spine. Additionally, forward head posture (FHP) alters the center of gravity (COG) of the body that lead to mechanical modifications related to postural control in the torso and every joint. The body attempts to adapt to these changes by altering its balance control mechanisms; these adaptations decrease balance ability while performing different activities and increase the risk of falling and musculoskeletal injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders aged 18-25 years old with forward head posture will be included in this study.
* Subjects have forward head posture if the craniovertebral angle ≤ 50.
* Subjects complain non- specific neck pain for at least 3 months or at least two episodes of non-specific neck pain during the last three months.
* Normal body mass index (18- 24.9).

Exclusion Criteria:

* Subjects with any spinal problems.
* Temporo-mandibular disease.
* Subjects with experience in Pilates and who will not sedentary were excluded from the study.
* Previous surgery in the neck and shoulder regions
* Current participation in a structured exercises program
* Neurological symptoms of the upper extremities during screening tests (e.g., Spurling test and upper limb tension tests)
* Red flags suggesting of cancer, infection, vascular insufficiency.
* Cervical radiculopathy or myelopathy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | up to twelve weeks
  will be measured by Biodex balance system
Craniovertebral angle | up to twelve weeks
  will be measured by photogrammetric method

SECONDARY OUTCOMES:
pain intensity | up to twelve weeks
  by visual analogue scale (VAS) 10 cm line with 2 ends, 0 and 10 ends 0 end means no pain 10 end means the worst pain
cervical range of motion | up to twelve weeks
  by cervical range of motion device (CROM)
Function of daily life | up to twelve weeks
  by Arabic version of neck disability index

CONTACTS AND LOCATIONS:
Overall Officials: Haytham M Elhafez, Professor, Study Director — professor of physical therapy- cairo university
Locations (1):
- Faculty of Physical Therapy-Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we will share the results of the trial 1-craniovertebral angle 2-dynamic balance 3-pain level of neck area 4-function of daily life 5-cervical range of motion
Supporting Information: Study Protocol
Time Frame: one year
Access Criteria: the criteria will be accessed by the publication of trials in international journal